CLINICAL TRIAL: NCT01257945
Title: Exercise, Physical Function, and Parkinson's Disease
Brief Title: Exercise for People With Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02-0750; R01HD043770 (NIH)
Record Dates: First submitted 2010-12-07; First posted 2010-12-10 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-10

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise; Pliability

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Flexibility & Function (Experimental): Subjects take part in an exercise program based on flexibility and function.
  Interventions: Behavioral: Flexibility and Function exercise program
- Aerobic Exercise (Experimental): Subjects will take part in an aerobic exercise program
  Interventions: Behavioral: Aerobic Exercise
- Home exercise (Other): Standard of care home exercise program
  Interventions: Behavioral: Home exercise program

INTERVENTIONS:
Behavioral: Aerobic Exercise
  Arms: Aerobic Exercise
Behavioral: Flexibility and Function exercise program
  Arms: Flexibility & Function
Behavioral: Home exercise program
  Arms: Home exercise

SUMMARY:
This randomized, controlled exercise intervention with three groups compares two exercise approaches to standard of care. Supervised interventions are administered for four months, with emphasis on patients adopting exercise habits to continue to exercise for an additional 12 months. Functional outcomes are measured at the completion of the supervised exercise (4 months) as well as 10 and 16 months.

DETAILED DESCRIPTION:
This randomized, controlled exercise intervention study compares physical therapy interventions for people in early and mid-stages of Parkinson's disease. Two different approaches to exercise are compared to standard of care. The two exercise programs consist of supervised interventions, administered for four months, with emphasis on patients adopting exercise habits to continue to exercise for an additional 12 months. The standard of care program consists of a home program in which participants exercise in a group setting once a month with an exercise trainer. Functional outcomes are measured at the completion of the supervised exercise at 4 months as well as 10 and 16 months. This study is the first long term exercise study for people with Parkinson's disease PD of which we are aware and is the most comprehensive examination of exercise for people with PD to date. Results of this study will provide definitive information regarding the best approach to exercise for people in early and mid stages of PD, both in terms of immediate 4 month and long term 16 month effects.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's Disease
* Hoehn & Yahr stages 1-3.5

Exclusion Criteria:

* Cardiovascular contraindications to aerobic exercise
* Reliance on walker or wheelchair
* Psychiatric conditions
* DBS or other surgeries
* Any other conditions that would interfere with exercise

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2003-04; Primary Completion 2010-04 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Functional Reach | baseline, 4, 10, 16 months
  Measure of balance

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Schenkman, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

REFERENCES:
- [Background] Christiansen CL, Schenkman ML, McFann K, Wolfe P, Kohrt WM. Walking economy in people with Parkinson's disease. Mov Disord. 2009 Jul 30;24(10):1481-7. doi: 10.1002/mds.22621. PMID 19441128
- [Result] Schenkman M, Hall D, Kumar R, Kohrt WM. Endurance exercise training to improve economy of movement of people with Parkinson disease: three case reports. Phys Ther. 2008 Jan;88(1):63-76. doi: 10.2522/ptj.20060351. Epub 2007 Oct 16. PMID 17940108
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886
- [Derived] Schenkman M, Hall DA, Baron AE, Schwartz RS, Mettler P, Kohrt WM. Exercise for people in early- or mid-stage Parkinson disease: a 16-month randomized controlled trial. Phys Ther. 2012 Nov;92(11):1395-410. doi: 10.2522/ptj.20110472. Epub 2012 Jul 19. PMID 22822237